CLINICAL TRIAL: NCT00523042
Title: Inhaled Preprandial Human Insulin With the AERx® iMS Versus Subcutaneous Injected Insulin Aspart in Subjects With Diabetes and Asthma: A 52-week, Open-label, Multinational, Randomised, Parallel Trial to Investigate Long-term Safety
Brief Title: Safety of Inhaled Preprandial Human Insulin in Subjects With Diabetes and Asthma
Acronym: iINHALE 9
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1616
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Asthma
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Asthma | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: inhaled human insulin
- B (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Treat-to-target dose titration scheme, injection s.c.
  Other Names: NovoRapid®; NovoLog®
  Arms: B
Drug: inhaled human insulin — Treat-to-target dose titration scheme, inhalation.
  Arms: A

SUMMARY:
This trial is conducted in Europe, Asia, Oceania and the United States of America (USA).

This is a one-year clinical trial to compare the safety of inhaled preprandial human insulin to subcutaneous insulin aspart in subjects with type 1 or 2 diabetes and asthma.

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* Treatment with insulin and/or oral anti-diabetic drugs
* Asthma for at least 6 months
* Positive airway reversibility/bronchoprovocation test or documented positive test in the last 3 years
* HbA1C less than or equal to 11.0 %
* Body Mass Index (BMI) less than or equal to 40.0 kg/m2

Exclusion Criteria:

* Current smoking or smoking within the last 6 months
* Other current acute or chronic pulmonary disease excluding asthma
* Recurrent severe hypoglycaemia
* Proliferative retinopathy or maculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08-30 (Actual); Primary Completion 2008-02-28 (Actual); Study Completion 2008-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in lung function, chest X-rays, or asthma exacerbation frequency | after 52 weeks of treatment

SECONDARY OUTCOMES:
Diabetes control measured by change in HbA1c | from baseline to end of treatment
Laboratory assessments (biochemistry, insulin antibodies, blood count) | from baseline to end of treatment
Preprandial insulin doses | for the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (31):
- United States (9):
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Spokane, Washington
- Australia (8):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Auchenflower
  - Novo Nordisk Investigational Site, Kippa-Ring
- India (6):
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Mumbai
  - Novo Nordisk Investigational Site, Pune
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Pulau Pinang
- Novo Nordisk Investigational Site, Belgrade, Serbia and Montenegro
- Slovakia (4):
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Ľubochňa
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Žilina

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com